CLINICAL TRIAL: NCT06903975
Title: The Effect of Injection of prabotulinumtoxinA-xvfs (Jeuveau) Into the Bilateral Sternocleidomastoid Muscles on Neck Circumference and Aesthetics
Brief Title: BoTox Into the Sternocleidomastoid Muscles (SCM)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Evolus, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-45473
Record Dates: First submitted 2025-03-26; First posted 2025-04-01 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Neck Muscle Issue
Keywords: Neck circumference; Neck aesthetics; Sternocleidomastoid muscles (SCM); Botulinum injection; PrabotulinumtoxinA-xvfs injection
MeSH Terms: interventions — prabotulinumtoxin A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Botulinum injection into SCM (Experimental): All participants will receive bilateral botulinum injections into the SCM.
  Interventions: Drug: prabotulinumtoxinA-xvfs

INTERVENTIONS:
Drug: prabotulinumtoxinA-xvfs — Each participant will receive 60 units (U) of prabotulinumtoxinA-xvfs into each SCM for a total of 120 U. Participants will return in 2 weeks to determine if any touch-up injection is needed.
  Other Names: Jeuveau

SUMMARY:
Botulinum toxin injections have been used both in the face and neck for many years. However, injection into the sternocleidomastoid muscle (SCM) has only been done to treat neck spasms. In this study botulinum toxin will be injected into the SCM to determine if this will result in a temporary slimming effect on the neck and produce a more feminine, youthful neck contour.

DETAILED DESCRIPTION:
The specific study objectives are to determine if:

* the neck circumference is decreased at 4 weeks after botulinum toxin (prabotulinumtoxinA-xvfs) injection.
* patients can appreciate a difference in their neck contour, self-confidence, and the way they perceive themselves post-injection via an aesthetics outcome and a neck perception survey.
* injection of the botulinum toxin into the sternocleidomastoid muscle is safe to perform based on adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age eligible individual seeking a more feminine neck appearance

Exclusion Criteria:

* Prior neuromodulator injections in the sternocleidomastoid muscles (SCM) within the past year
* Current anticoagulant use
* Body mass index (BMI) >30
* Anticipation of significant weight gain or loss during the study period (e.g. patients taking or planning to take within the study period a semaglutide medication.)
* Prior allergy to botulinum toxin A
* Currently pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Neck circumference | Baseline, 4 weeks
  A standard tape measure will be used and circumference recorded in centimeters

SECONDARY OUTCOMES:
Post injection neck appearance | 4 weeks
  A 5-item investigator developed questionnaire will be used to assess each participant's opinion about their neck appearance after the botulinum toxin injections. Each item has 4 potential responses from 1=Definitely disagree to 4=Definitely agree. Total scores can range from 5 to 20 and higher scores suggest more positive opinions about their neck appearance.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Spiegel, MD, Principal Investigator — Boston Medical Center and The Spiegel Center
Locations (1):
- The Spiegel Center, Newton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No